CLINICAL TRIAL: NCT06462560
Title: Improving Physical Function and Quality of Life in Adults With Knee Osteoarthritis Utilizing an Online Live and Interactive Fitness Training Program (Vivo Knee OA)
Brief Title: Live and Interactive Fitness Training Program (Vivo Knee OA)
Acronym: LIFT-OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Impactiv, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1052693
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vivo Online Exercise program (Experimental)
  Interventions: Other: Vivo Online Exercise Program
- Medbridge Home Exercise Program (Active Comparator)
  Interventions: Other: Medbridge Home program

INTERVENTIONS:
Other: Vivo Online Exercise Program — Virtual online exercise programs conducted by the Vivo team consisting of multiple time a week group live programs
  Arms: Vivo Online Exercise program
Other: Medbridge Home program — At home exercise program accessed through exercise descriptions and short vidoes
  Arms: Medbridge Home Exercise Program

SUMMARY:
Potential participants will be screened at clinic. Patients who meet eligibility criteria will be considered for study. After written informed consent is obtained, participants will complete baseline testing and participants who meet eligibility criteria will be randomized 1:1 to 2 treatment arms: Vivo Arm: Vivo twice a week for 6 months and Usual Care Arm: meet with ATC and given Medbridge home exercise program for 6 months. All participants will be followed for 12 months, and will be assessed at 3-,6-, and 12-months. All participants will complete functional assessments, OA patient reported outcomes measures, quality of life, exercise self-efficacy, and fall risk questionnaires, and health care utilization report at each testing visit. A subset of Vivo participants will be asked satisfaction questions at the 3 and 6 month time points.

ELIGIBILITY:
Inclusion Criteria:

* 55-85 years of age
* Diagnosis of Osteoarthritis within the prior 6 months
* Symptomatic OA defined as self-report:

  * Pain in the knee(s) on most days of the month
  * Difficulty with at least one of the following because of knee pain:

    * walking ¼ of a mile
    * climbing stairs
    * getting in and out of a car, bath, or bed
    * rising from a chair
    * or performing shopping, cleaning, or self-care activities
* Radiographic KL grade II-III (using Kellgren and Lawrence criteria) of one or both knees
* Physically able to participate in strength training - able to do one chair stand unassisted in order to test change in 30-second chair stand
* Ambulatory and community-dwelling
* Sedentary or insufficiently active as measured by the PAVS
* Access to Wi-Fi in defined exercise space
* BMI of 20-34.9 kg/m2
* Document medication specific to OA and knee pain
* Willing and able to provide consent

Exclusion Criteria:

* Neurological conditions causing functional impairments (Parkinson's disease, MS, ALS)
* Diagnosis of dementia
* Inability to complete ≥1 ADLs without assistance.
* Knee surgery in the past 6 months
* Severe osteoporosis T-score < -3.5
* No concurrent enrollment in physical therapy for knee pain
* No concurrent enrollment in the Intermountain Arthrofit program
* Under the age of 55 or ≥85
* Asymptomatic OA
* Not having knee pain or having significant knee pain (WOMAC Pain score of ≤3 or ≥18)
* KL Grade 1 or 4
* BMI above 34.9 kg/m2 or ≤20 kg/m2
* Participation in formal strength training more than 30 minutes a week in the past 6 months.
* PAVS - Participating in 150 minutes per week of moderate intensity physical activity or 75 minutes of vigorous intensity activity, or an equivalent combination of moderate and vigorous intensity physical activity.
* Co-morbid disease that would threaten safety or impair ability to participate in a live and interactive strength training program
* Symptomatic or severe coronary artery disease; peripheral vascular disease
* Untreated hypertension
* Active cancer other than skin cancer

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2024-04-28 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint 1 | 6 months post intervention
  Changes from baseline in number of chair stands done in 30-seconds at 3 and 6 months.

SECONDARY OUTCOMES:
Secondary Endpoint 1 | 6 months post intervention
  Changes from baseline in WOMAC score at 3 and 6 months.
Secondary Endpoint 2 | 6 months post intervention
  Changes from baseline in length of time (seconds) to do 1-leg balance stance at 3 and 6 months.
Secondary Endpoint 3 | 6 months post intervention
  Changes from baseline in seconds to complete the 8-foot up and go at 3 and 6 months.
Secondary Endpoint 4 | 6 months post intervention
  Changes from baseline in number of knee raises completed in 2-minute knee raise at 3 and 6 months
Secondary Endpoint 5 | 6 months post intervention
  Changes from baseline in number of arm-curls done in 30 seconds at 3 and 6 months
Secondary Endpoint 6 | 6 months post intervention
  Changes from baseline in PROMIS-Plus-Osteoarthritis of the Knee (OAK) score at 3 and 6 months
Secondary Endpoint 7 | 6 months post intervention
  Changes from baseline in exercise self-efficacy scale score at 3 and 6 months
Secondary Endpoint 8 | 6 months post intervention
  Changes from baseline in quality of life (SF-36 score) at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Beutler, MD, Principal Investigator — Intermountain Health
Locations (1):
- Intermountain Health, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No